CLINICAL TRIAL: NCT04502121
Title: Preoperative Optimization of Cardiac Valve Patients' Expectations - a Randomized Controlled Trial
Brief Title: Preoperative Optimization of Cardiac Valve Patients' Expectations
Acronym: ValvEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Heart Centre Rotenburg (Other); Justus-Liebig University Gießen Medical Center (Unknown)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ValvEx
Record Dates: First submitted 2020-06-23; First posted 2020-08-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Valve Disease
Keywords: Expectations; Preoperative intervention; placebo effect; cardiac valve surgery; clinical trial; recovery
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to the intervention group (IG) or the control group (SOC). The intervention group will receive a psychological preoperative intervention to optimize expectations (in addition to standard medical care). The control group will receive the standard of care only.
Who Masked: Care Provider
Masking Description: The psychologist will inform the patient about the group s/he is randomly assigned to. The medical staff will not receive any information about the group a patient is allocated to and therefore be masked regarding group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental)
  Interventions: Behavioral: EXPECT: Preoperative optimization of cardiac valve patient's expectations
- Standard of Care (SOC) (No Intervention)

INTERVENTIONS:
Behavioral: EXPECT: Preoperative optimization of cardiac valve patient's expectations — The psychological, preoperative intervention follows a treatment manual. Patients get a personal intervention one day before surgery (30-40 minutes). It includes the development of an individual, subjectively perceived disease model, the treatment outcome expectations and the personalized outcome expectancy. Additionally they get two booster telephone calls 4 and 8 weeks after the surgery to recall the discussed topics and to talk about their recovery process (10-15 minutes).
  Arms: Intervention group (IG)

SUMMARY:
Recovery after surgery depends on psychological factors such as preoperative information, expectations and surgery-associated anxiety. Prior studies have shown that even short preoperative psychological interventions can improve postoperative outcomes in heart surgery patients. However, what content works best for which patient group and how long an intervention has to be is still largely unknown. The aims of this study are thus to examine if the developed preoperative psychological intervention (i) reduces preoperative anxiety, (ii) increases positive expectations, and (iii) improves the long-term outcome postoperative recovery. Therefore, a brief intervention has been developed. Heart valve patients who undergo a heart surgery will be randomized into two groups (Control vs. intervention group) after baseline assessment. Following this the intervention group will participate in the psychological intervention (30-40 minutes). To increase patients' positive expectations the intervention will focus on treatment outcome expectations and personal control expectations. Furthermore, patients in the intervention group will have two booster-telephone calls (four and eight weeks after the surgery) to check if their developed plans work out. The control group will receive the standard medical procedure. Both groups will fill out questionnaires again at the evening before the surgery, around one week after the surgery and three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective cardiac valve procedure
* Age 18 or above
* Fluency in German
* Informed consent

Exclusion Criteria:

* Comorbid medical/psychiatric condition that causes more extensive disability than the coronary condition
* Participation in other research programs: in agreement with Coordinating Investigator patient can participate substudies, if this do not interfere with the main study
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain Disability Index (PDI) from Baseline to one day pre-surgery to one week post-surgery to three months post-surgery | Baseline, one day pre-surgery, up to one week post-surgery, up to three months post-surgery
  Items range from 0 (no disability at all) - 10 (total disability). Consequently higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 0 (no restriction), 1 (nearly not restricted) - 5 (very strongly restricted). Consequently higher scores mean a worse outcome.
Change in Health Related Quality of Life (Short Form 12, SF-12) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  There are different item scales. The item scale of the first item (General health perceptions) ranges from 1 (excellent) to 5 (bad). The item scales of the second and third item (limitations in physical activities because of health problems) range from 1 (yes, absolutely restricted) to 2 (yes, a bit restricted) to 3 (no, not restricted at all). The item scales of the items 4-7 (limitations in usual role activities because of physical health or emotional problems) are just "yes" and "no". The item scale of the eighth item (bodily pain) ranges from 1 (Absolutely not) to 5 (a lot). The item scales of the items 9-12 (general mental health, vitality and limitations in social activities because of physical or emotional problems) range from 1 (always) to 5 (never).
Change in Patient health questionnaire screener (PHQ) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (not at all) - 4 (nearly everyday). Consequently higher scores mean a worse outcome.
Change in Generalized Anxiety Disorder 7 (GAD-7) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (not at all) - 4 (nearly everyday). Consequently higher scores mean a worse outcome.
Change in Anxiety (The Amsterdam Preoperative Anxiety and Information Scale, APAIS) from Baseline to one day pre-surgery | Baseline, one day pre-surgery
  Items range from 1 (not at all) - 5 (extremely). Higher scores mean patients are more interested in information and do have greater worries.
Days the patient stays in the hospital, days at the intensive care unit | up to one week post-surgery
Change of Concentration of Inflammatory marker C-reactive protein (CRP) in mg/l | Baseline, up to one day, two days and five days post-surgery
  Change from baseline to postoperative day 1 (POD1) to approx. POD2 to approx. POD 5; higher scores mean a worse outcome.

OTHER OUTCOMES:
Change in The Primary Appraisal Secondary Appraisal questionnaire (PASA) from Baseline to one day pre-surgery to one week post-surgery | Baseline, one day pre-surgery, up to one week post-surgery
  Items range from 0 (absolutely wrong) - 6 (absolutely right). Higher scores mean a better outcome.
Change in Patients' Illness Perception (Brief Illness Perception Questionnaire, B-IPQ) from Baseline to 1 week post-surgery to 3 months after surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  The B-IPQ surveys the cognitive and emotional representations of illness. Item 1-5 measure cognitive illness representations (consequences, timeline, personal control, treatment control, andidentity). Item 6 and 8 quantify emotional representations (concern & emotions). Item 7 assesses illness comprehensibility. Item 9 is an open question (three most important causal factors in their illness). Items range from 0-10: item 1: no disability at all to very strong disability, item 2: really short to forever, item 3: no control at all zo extreme control, item 4: not at all to extremely helpful, item 5: no complaints at all to very much and strong complaints, item 6: no worries at all to extreme worries, item 7: not at all to very clear, item 8: emotionally not included at all to emotional extremely included.
Change in patients' expectations (Expected Illness Perception Questionnaire, IPQ-E) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (absolutely wrong) - 5 (absolutely right). Higher scores mean a better outcome.
Change in patients optimism (Life-Orientation-Test Revised, LOT-R) from Baseline to one week post-surgery to three months post-surgery | Baseline, up to one week post-surgery, up to three months post-surgery
  Items range from 1 (absolutely) - 5 (absolutely not). Higher scores mean a worse outcome.
Personality (Big Five Inventory, BFI-10) | Baseline
  Items range from 1 (disagree strongly) - 5 (agree strongly). The questionnaire includes the scales "openness to experience", "conscientiousness", "extraversion", agreeableness and neuroticism.
Patients' experience with prior surgeries | Baseline
  Rating of experience with own prior surgeries. Rating of experience with surgeries of close others. First patients are asked if they or close others had a prior surgery before (yes/no). If they answer yes, they are asked to rate their or their close others experience (item ranges from 1 (very bad) - 5 (very good).
Surgery procedure (planned and realized) | Baseline, up to one week post-surgery
  The planned and the realized surgical approach (minimally invasive or open) will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Clinical Psychology and Psychotherapy Dept. of Psychology, Philipps-University Marburg; Ardawan Rastan, Prof. Dr., Principal Investigator — Cardiac surgery University Hospital Gießen und Marburg
Locations (1):
- UKGM Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Auer CJ, Glombiewski JA, Doering BK, Winkler A, Laferton JA, Broadbent E, Rief W. Patients' Expectations Predict Surgery Outcomes: A Meta-Analysis. Int J Behav Med. 2016 Feb;23(1):49-62. doi: 10.1007/s12529-015-9500-4. PMID 26223485
- [Background] Juergens MC, Seekatz B, Moosdorf RG, Petrie KJ, Rief W. Illness beliefs before cardiac surgery predict disability, quality of life, and depression 3 months later. J Psychosom Res. 2010 Jun;68(6):553-60. doi: 10.1016/j.jpsychores.2009.10.004. Epub 2009 Dec 5. PMID 20488272
- [Background] Laferton JA, Kube T, Salzmann S, Auer CJ, Shedden-Mora MC. Patients' Expectations Regarding Medical Treatment: A Critical Review of Concepts and Their Assessment. Front Psychol. 2017 Feb 21;8:233. doi: 10.3389/fpsyg.2017.00233. eCollection 2017. PMID 28270786
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Rief W, Shedden-Mora MC, Laferton JA, Auer C, Petrie KJ, Salzmann S, Schedlowski M, Moosdorf R. Preoperative optimization of patient expectations improves long-term outcome in heart surgery patients: results of the randomized controlled PSY-HEART trial. BMC Med. 2017 Jan 10;15(1):4. doi: 10.1186/s12916-016-0767-3. PMID 28069021
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Löwe, B., Spitzer, R. L., Zipfel, S., & Herzog, W. (2002). PHQ-D Gesundheitsfragebogen für Patienten (German Version of the Patient Health Questionnaire). Karlsruhe: Pfizer.
- [Background] Rector TS, Kubo SH, Cohn JN. Validity of the Minnesota Living with Heart Failure questionnaire as a measure of therapeutic response to enalapril or placebo. Am J Cardiol. 1993 May 1;71(12):1106-7. doi: 10.1016/0002-9149(93)90582-w. No abstract available. PMID 8475878
- [Background] Rief, W., & Glombiewski, J. A. (2016). Erwartungsfokussierte Psychotherapeutische Interventionen (EFPI). Verhaltenstherapie, 26(1), 47-54.
- [Background] Salzmann, S., Laferton, J., Auer, C., Shedden-Mora, M., Wambach, K., & Rief, W. (2018). Patientenerwartungen optimieren: Beschreibung einer präoperativen Kurzintervention am Beispiel von Patienten vor einer Bypass-Operation. Verhaltenstherapie, 28(3), 157-165.
- [Background] Gaab, J. (2009). PASA-Primary Appraisal Secondary Appraisal-Ein Fragebogen zur Erfassung von situations-bezogenen kognitiven Bewertungen. Verhaltenstherapie, 19(2), 114-115.
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Rammstedt, B. und O. P. John, 2007: Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. Journal of Research in Personality 41: 203-212
- [Derived] Horn N, Gartner L, Rastan AJ, Andrasi TB, Lenz J, Boning A, Salzmann-Djufri M, Puvogel U, Niemann B, Genovese M, Habash S, Euteneuer F, Rief W, Salzmann S. Effects of a preoperative psychological expectation-focused intervention in patients undergoing valvular surgery - the randomized controlled ValvEx (valve patients' expectations) study. Am Heart J. 2025 Apr;282:156-169. doi: 10.1016/j.ahj.2025.01.006. Epub 2025 Jan 17. PMID 39827935
- [Derived] Horn N, Gartner L, Rastan AJ, Andrasi TB, Lenz J, Boning A, Salzmann-Djufri M, Puvogel U, Genovese M, Kus S, Rief W, Salzmann S. Preoperative optimization of cardiac valve patients' expectations: Study protocol of the randomized controlled ValvEx-trial. Front Cardiovasc Med. 2023 Mar 2;10:1105507. doi: 10.3389/fcvm.2023.1105507. eCollection 2023. PMID 36937912